CLINICAL TRIAL: NCT02886884
Title: A Phase I/II, Randomized, Double Blind, Pilot Trial to Evaluate the Safety and Efficacy of Allogeneic Mesenchymal Human Stem Cells Infusion Therapy for Endothelial DySfunctiOn in Diabetic Subjects
Brief Title: Allogeneic Mesenchymal Human Stem Cells Infusion Therapy for Endothelial DySfunctiOn in Diabetic Subjects
Acronym: ACESO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joshua M Hare (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Sponsor - Investigator, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20160686; 1R01HL134558-01 (NIH)
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Results first posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Endothelial dysfunction; Stem cells
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pilot phase is open label. Randomized phase is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pilot Phase 20 million allogeneic hMSCs (Experimental): Participants in this group will receive one peripheral intravenous infusion of 20 million allogeneic Mesenchymal Human Stem Cells (hMSCs)
  Interventions: Drug: 20 million Allogeneic Mesenchymal Human Stem Cells
- Pilot Phase 100 million hMSCs (Experimental): Participants in this group will receive one peripheral intravenous infusion of 100 million allogeneic Mesenchymal Human Stem Cells (hMSCs)
  Interventions: Drug: 100 million Allogeneic Mesenchymal Human Stem Cells
- Randomized Phase 20 million allogeneic hMSCs (Experimental): Participants in this group will receive one peripheral intravenous infusion of 20 million allogeneic Mesenchymal Human Stem Cells (hMSCs)
  Interventions: Drug: 20 million Allogeneic Mesenchymal Human Stem Cells
- Randomized Phase 100 million allogeneic hMSCs (Experimental): Participants in this group will receive one peripheral intravenous infusion of 100 million allogeneic Mesenchymal Human Stem Cells (hMSCs)
  Interventions: Drug: 100 million Allogeneic Mesenchymal Human Stem Cells

INTERVENTIONS:
Drug: 20 million Allogeneic Mesenchymal Human Stem Cells — 1 single intravenous infusion
  Other Names: allo-hMSCs; stem cells
  Arms: Pilot Phase 20 million allogeneic hMSCs; Randomized Phase 20 million allogeneic hMSCs
Drug: 100 million Allogeneic Mesenchymal Human Stem Cells — 1 single intravenous infusion
  Other Names: allo-hMSCs; stem cells
  Arms: Pilot Phase 100 million hMSCs; Randomized Phase 100 million allogeneic hMSCs

SUMMARY:
This is a 16 subject trial to demonstrate the safety of allogeneic hMSCs administered via infusion therapy for diabetic subjects with endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 21 and < 90 (inclusive) years of age.
* Provide written informed consent.
* Have endothelial dysfunction defined by impaired flow-mediated vasodilation (FMD <7%).
* Have an ejection fraction > 45% by gated blood pool scan, two- dimensional echocardiogram, cardiac MRI, cardiac CT or left ventriculogram within the prior 3 months.
* Have Diabetes mellitus type 2 documented by hemoglobin adult type 1 component (A1C) > 7% or on medical therapy for diabetes.
* Females of childbearing potential must use two forms of birth control for the duration of the study. Female subjects must undergo a blood or urine pregnancy test at screening and within 36 hours prior to infusion.

Exclusion Criteria:

In order to participate in this study, a subject Must Not:

* Be younger than 21 years or older than 90 years of age.
* Have a baseline glomerular filtration rate <35 ml/min 1.73m^2 estimated using the Modification of Diet in renal disease (MDRD) formula.
* Have an ejection fraction <45% by gated blood pool scan, two-dimensional echocardiogram, cardiac MRI, cardiac CT or left ventriculogram within the past year, as documented by medical history.
* Have poorly controlled blood glucose levels with hemoglobin A1C > 8.5%.
* Have a history of proliferative retinopathy or severe neuropathy requiring medical treatment.
* Have a hematologic abnormality as evidenced by hematocrit < 25%, white blood cell < 2,500/ul or platelet values < 100,000/ul without another explanation.
* Have liver dysfunction, as evidenced by enzymes (AST and ALT) greater than three times the upper limit of normal.
* Have a bleeding diathesis or coagulopathy (INR > 1.3), cannot be withdrawn from anticoagulation therapy, or will refuse blood transfusions.
* Have Lymphadenectomy or Lymph node dissection in the right arm.
* Be an organ transplant recipient or have a history of organ or cell transplant rejection.
* Have a clinical history of malignancy within the past 5 years (i.e., subjects with prior malignancy must be disease free for 5 years), except curatively- treated basal cell or squamous cell carcinoma, or cervical carcinoma.
* Have a condition that limits lifespan to < 1 year.
* Have a history of drug or alcohol abuse within the past 24 months.
* Be on chronic therapy with immunosuppressant medication, such as corticosteroids or Tumor Necrosis Factor - alpha (TNFα) antagonists.
* Be serum positive for HIV, Syphilis - VDRL (Confirmation with FTA-ABS if needed (Syphilis)), hepatitis B surface antigen or viremic hepatitis C.
* Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.
* Be pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods.
* Any other condition that in the judgment of the Investigator would be a contraindication to enrollment or follow-up.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Hare, MD, Principal Investigator — ISCI / University of Miami Miller School of Medicine
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Interdisciplinary stem cell institute at the University of Miami website — http://isci.med.miami.edu

RESULTS

PARTICIPANT FLOW:
Period: Treatment
Arm/Group | Pilot Phase 20 Million Allogeneic hMSCs | Pilot Phase 100 Million hMSCs | Randomized Phase 20 Million Allogeneic hMSCs | Randomized Phase 100 Million Allogeneic hMSCs
Started | 3 | 3 | 5 | 5
Completed | 3 | 3 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Follow-up
Arm/Group | Pilot Phase 20 Million Allogeneic hMSCs | Pilot Phase 100 Million hMSCs | Randomized Phase 20 Million Allogeneic hMSCs | Randomized Phase 100 Million Allogeneic hMSCs
Started | 3 | 3 | 5 | 5
Completed | 3 | 3 | 5 | 4
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot Phase 20 Million Allogeneic hMSCs | Pilot Phase 100 Million hMSCs | Randomized Phase 20 Million Allogeneic hMSCs | Randomized Phase 100 Million Allogeneic hMSCs | Total
Number analyzed (Participants) | 3 | 3 | 5 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (13.6) | 69.3 (6.7) | 59.8 (13.7) | 62.0 (8.1) | 64.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 3 | 2 | 5
  Male | 3 | 3 | 2 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 2 | 5
  Not Hispanic or Latino | 3 | 3 | 2 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 2 | 3
  White | 2 | 3 | 4 | 3 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Serious Adverse Events (TE-SAEs)
Description: TE-SAEs as evaluated by the investigator which may include but not limited to: death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities.
Time Frame: Up to one month (post infusion)
Measure: Number; unit: Treatment Emergent SAE
Arm/Group | Pilot Phase 20 Million Allogeneic hMSCs | Pilot Phase 100 Million hMSCs | Randomized Phase 20 Million Allogeneic hMSCs | Randomized Phase 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 3 | 3 | 5 | 5
Treatment Emergent SAE | 0 | 0 | 0 | 0

2. Secondary Outcome: EPC-CFU Levels
Description: Endothelial Progenitor Cell Colony Forming Units (EPC-CFU) will be assessed from blood samples
Time Frame: At Baseline, Day 3, Day 7, Day 14, Day 28, Day 90, Day 180, Day 365
Population: Not all participants completed required blood draw at each timepoint.
Measure: Mean (Standard Deviation); unit: Colony forming units
Arm/Group | Pilot Phase 20 Million Allogeneic hMSCs | Pilot Phase 100 Million hMSCs | Randomized Phase 20 Million Allogeneic hMSCs | Randomized Phase 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 3 | 3 | 5 | 5
Colony forming units
  Baseline | 2.06 (1.35) | 3.16 (1.92) | 2.37 (2.60) | 1.93 (1.38)
  Day 3 | 3.39 (3.31) | 5.50 (3.01) | 4.37 (3.20) | 2.80 (1.72)
  Day 7 | 9.28 (14.21) | 6.94 (8.67) | 6.07 (3.51) | 5.53 (4.78)
  Day 14 | 6.11 (8.74) | 19.72 (17.49) | 8.23 (4.07) | 11.70 (11.58)
  Day 28 | 7.83 (5.20) | 21.83 (2.96) | 2.50 (0.96) | 6.70 (8.27)
  Day 90: number analyzed (Participants) | 2 | 3 | 5 | 5
  Day 90 | 9.17 (8.72) | 14.17 (2.32) | 1.90 (2.50) | 6.50 (8.16)
  Day 180 | 8.39 (7.07) | 14.33 (3.12) | 2.45 (3.41) | 4.50 (6.46)
  Day 365: number analyzed (Participants) | 3 | 3 | 4 | 3
  Day 365 | 6.89 (4.68) | 8.83 (3.91) | 1.04 (0.63) | 2.94 (4.25)

3. Secondary Outcome: CRP Marker Levels
Description: C-Reactive Protein (CRP) levels will be assessed from blood samples and reported in mg/L
Time Frame: At Baseline, Day 3, Day 7, Day 14, Day 28, Day 90, Day 180, Day 365
Population: Blood samples were collected. However, due to cost and logistical reasons, the samples were not analyzed and hence no data were generated
Arm/Group | Pilot Phase 20 Million Allogeneic hMSCs | Pilot Phase 100 Million hMSCs | Randomized Phase 20 Million Allogeneic hMSCs | Randomized Phase 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Circulating Angiogenic Factor Levels
Description: Circulating Angiogenic Factor levels including Vascular Endothelial Growth Factor (VEGF), Stem Cell Factor (SCF) and Stromal Cell-Derived Factor 1 (SDF-1) will be assessed from blood samples and reported in ng/mL
Time Frame: At Baseline, Day 3, Day 7, Day 14, Day 28, Day 90, Day 180, Day 365
Population: as for outcome 3
Arm/Group | Pilot Phase 20 Million Allogeneic hMSCs | Pilot Phase 100 Million hMSCs | Randomized Phase 20 Million Allogeneic hMSCs | Randomized Phase 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Flow Mediated Diameter Percentage (FMD%)
Description: FMD will be assessed using brachial artery ultrasound
Time Frame: At Baseline, Day 3, Day 7, Day 14, Day 28, Day 90, Day 180, Day 365
Population: Not all participants completed the brachial artery ultrasound at each timepoint.
Measure: Mean (Standard Deviation); unit: Percent dilation of brachial artery
Arm/Group | Pilot Phase 20 Million Allogeneic hMSCs | Pilot Phase 100 Million hMSCs | Randomized Phase 20 Million Allogeneic hMSCs | Randomized Phase 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 3 | 3 | 5 | 5
Percent dilation of brachial artery
  Baseline | 2.55 (1.11) | 4.33 (2.61) | 4.55 (1.17) | 3.11 (1.92)
  Day 3 | 2.86 (1.96) | 4.76 (1.46) | 5.19 (1.33) | 4.99 (1.98)
  Day 7 | 2.97 (1.61) | 5.06 (3.70) | 4.80 (0.98) | 5.35 (2.45)
  Day 14 | 2.62 (0.53) | 5.18 (3.78) | 5.10 (1.55) | 4.94 (1.50)
  Day 28 | 2.33 (1.35) | 4.45 (3.94) | 5.67 (2.63) | 6.19 (2.53)
  Day 90: number analyzed (Participants) | 2 | 3 | 5 | 5
  Day 90 | 1.26 (0.50) | 4.78 (2.49) | 5.65 (2.89) | 5.34 (2.44)
  Day 180 | 2.90 (1.74) | 4.32 (2.47) | 5.78 (3.11) | 4.04 (1.84)
  Day 365: number analyzed (Participants) | 3 | 3 | 4 | 3
  Day 365 | 1.81 (0.24) | 4.14 (0.38) | 3.88 (1.61) | 3.65 (1.75)

6. Secondary Outcome: Circulating Inflammatory Marker Levels
Description: Circulating inflammatory marker levels including Interleukin (IL) -1 and IL-6 will be assessed from blood samples and reported in pg/mL
Time Frame: At Baseline, Day 3, Day 7, Day 14, Day 28, Day 90, Day 180, Day 365
Population: as for outcome 3
Arm/Group | Pilot Phase 20 Million Allogeneic hMSCs | Pilot Phase 100 Million hMSCs | Randomized Phase 20 Million Allogeneic hMSCs | Randomized Phase 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Tumor Necrosis Factor (TNF) Alpha Levels
Description: Measured from blood samples (pg/mL)
Time Frame: At Baseline, Day 3, Day 7, Day 14, Day 28, Day 90, Day 180, Day 365
Population: Not all participants completed required blood draw at each timepoint.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pilot Phase 20 Million Allogeneic hMSCs | Pilot Phase 100 Million hMSCs | Randomized Phase 20 Million Allogeneic hMSCs | Randomized Phase 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 3 | 3 | 5 | 5
pg/mL
  Baseline: number analyzed (Participants) | 3 | 2 | 5 | 5
  Baseline | 0.79 (0.13) | 0.80 (0.19) | 0.85 (0.21) | 0.80 (0.12)
  Day 3: number analyzed (Participants) | 2 | 2 | 5 | 5
  Day 3 | 0.74 (0.04) | 0.86 (0.33) | 1.01 (0.24) | 0.81 (0.15)
  Day 7: number analyzed (Participants) | 2 | 3 | 5 | 5
  Day 7 | 0.77 (0.03) | 0.74 (0.09) | 0.90 (0.45) | 1.09 (0.55)
  Day 14 | 0.80 (0.04) | 1.01 (0.20) | 0.93 (0.41) | 0.90 (0.33)
  Day 28 | 0.69 (0.20) | 0.84 (0.17) | 0.84 (0.31) | 0.82 (0.19)
  Day 90: number analyzed (Participants) | 2 | 3 | 5 | 5
  Day 90 | 0.68 (0.15) | 0.81 (0.13) | 0.83 (0.10) | 0.71 (0.12)
  Day 180: number analyzed (Participants) | 1 | 3 | 5 | 5
  Day 180 | 17.10 (NA) — There is only one participant analyzed. Standard Deviation cannot be calculated. | 0.98 (0.51) | 0.79 (0.25) | 0.76 (0.10)
  Day 365: number analyzed (Participants) | 3 | 3 | 4 | 3
  Day 365 | 0.83 (0.23) | 0.95 (0.32) | 0.76 (0.08) | 0.81 (0.23)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Pilot Phase 20 Million Allogeneic hMSCs | Pilot Phase 100 Million hMSCs | Randomized Phase 20 Million Allogeneic hMSCs | Randomized Phase 100 Million Allogeneic hMSCs
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/5 | 1/5
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Phase 20 Million Allogeneic hMSCs (N=3) | Pilot Phase 100 Million hMSCs (N=3) | Randomized Phase 20 Million Allogeneic hMSCs (N=5) | Randomized Phase 100 Million Allogeneic hMSCs (N=5)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Removal of left lung nodule
Gastrointestinal Stromal Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Surgical Site Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Phase 20 Million Allogeneic hMSCs (N=3) | Pilot Phase 100 Million hMSCs (N=3) | Randomized Phase 20 Million Allogeneic hMSCs (N=5) | Randomized Phase 100 Million Allogeneic hMSCs (N=5)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated White Blood Cells with Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incomplete Right bundle branch block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal Edema, Deterioration of vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophogeal Reflux Disease Exacerbation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Recurrence of Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic Reaction to Flu shot (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mild allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital Herpes Simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Viral Illness (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Poor Diabetes Control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left Distal fibula fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal Urinalysis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinurea (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical Intraepithelial Neoplasia 1, Mild Dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bullous Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT02886884/Prot_SAP_000.pdf